CLINICAL TRIAL: NCT03122977
Title: Acute-phase Response Following Full-mouth Versus Quadrant Non-surgical Periodontal Treatment in Obese Subjects: A Randomized Clinical Trial
Brief Title: Acute-phase Response & Periodontal Treatment in Obese Patients
Acronym: PERIO-OBESE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Professor of Periodontology, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3399/11_B
Record Dates: First submitted 2017-03-08; First posted 2017-04-21 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Periodontal Diseases; Obesity
MeSH Terms: conditions — Periodontal Diseases; Obesity | interventions — Root Planing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full mouth scaling and root planing (Experimental): FM-SRP Non surgical periodontal treatment will be performed in all dentition within 24 hours
  Interventions: Procedure: FM-SRP
- Quadrant scaling and root planing (Active Comparator): Q-SRP Non surgical periodontal treatment will be performed in all dentition subdivided in four appointments. Each appointment will be performed in one week interval. In each appointment only a "quadrant" of the dentition will be instrumented.
  Interventions: Procedure: Q-SRP

INTERVENTIONS:
Procedure: FM-SRP — Supra- and sub-gingival mechanical instrumentation of the root surface of the whole dentition within 24 hours.
  Other Names: Full mouth scaling and root planing
  Arms: Full mouth scaling and root planing
Procedure: Q-SRP — Supra- and sub-gingival mechanical instrumentation of the root surface will be performed in all dentition subdivided in four appointments. Each appointment will be performed in one week interval. In each appointment only a "quadrant" of the dentition will be instrumented.
  Other Names: Quadrant scaling and root planing
  Arms: Quadrant scaling and root planing

SUMMARY:
The aim of this study is to compare quadrant scaling and root planing (Q-SRP) versus full-mouth treatment (FM-SRP) in terms of acute-phase responses following no surgical periodontal treatment in obese patients affected by periodontitis.

DETAILED DESCRIPTION:
Periodontal treatment, consisting in both supra- and sub-gingival mechanical instrumentation of the root surface (scaling and root planing), will be performed by a single periodontist on obese patients with periodontitis.

The aim of this study is to compare quadrant scaling and root planing (Q-SRP) versus full-mouth treatment (FM-SRP) in terms of acute-phase responses following non surgical periodontal treatment.

Treatment will be provided using both hand and ultrasonic instrumentation with ﬁne tips.

FM-SRP patients will received treatment within 24 h. Q-SRP patients will received four quadrants sessions of periodontal treatment with an interval of 1 week between sessions.

Vital, endothelial function and blood inflammatory parameters will be evaluated at baseline, 24 hours after the first treatment and after 3 months. Periodontal parameters will be evaluated at baseline and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Periodontal Disease
* 20% of periodontal pockets of the entire dentition
* 20% bleeding on probing of the entire dentition
* documented radiographic bone loss
* diagnosis of Obesity as measured through Body Mass Index (BMI) superior than 30

Exclusion Criteria:

* age younger than 18 years and older than 80 years
* pregnant or lactating females
* need of antibiotic coverage for periodontal treatment
* treatment with statin and/or acetylsalicylic acid
* BMI > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Levels C-Reactive Protein | Baseline, 24 hours and 3 months after treatment
  Changes in C reactive protein (CRP). Unit of measure: mg/L

SECONDARY OUTCOMES:
Full Mouth Plaque Score (FMPS) | Baseline and 3 months after treatment
  Changes in FMPS. Unit of Measure: %
Full Mouth Bleeding Score (FMBS) | Baseline and 3 months after treatment
  Changes in FMBS. Unit of Measure: %
Pocket probing depth (PPD) | Baseline and 3 months after treatment
  Changes in PPD. Unit of Measure: mm
Clinical attachment level (CAL) | Baseline and 3 months after treatment
  Changes in CAL. Unit of Measure: mm
Recession of the gingival margin (REC) | Baseline and 3 months after treatment
  Changes in REC. Unit of Measure: mm
Triglycerides | Baseline, 24 hours and 3 months after treatment
  Changes in triglycerides. Unit of measure: mmol/L
Low-density lipoprotein (LDL) | Baseline, 24 hours and 3 months after treatment
  Changes in LDL. Unit of measure: mmol/L
High-density lipoprotein (HDL) | Baseline, 24 hours and 3 months after treatment
  Changes in HDL. Unit of measure: mmol/L
Cholesterol | Baseline, 24 hours and 3 months after treatment
  Changes in total cholesterol. Unit of measure: mmol/L
Glycaemia | Baseline, 24 hours and 3 months after treatment
  Changes in blood glucose level; Unit of measure: mg/dL
Glycated Hemoglobin | Baseline and 3 months after treatment
  Changes in Glycated Hemoglobin level; Unit of measure: mmol/mol
Insulin | Baseline, 24 hours and 3 months after treatment
  Changes in Insulin level; Unit of measure: μU/mL
Systolic Blood Pressure (SBP) | Baseline, 24 hours and 3 months after treatment
  Changes in SBP; Unit of measure: mmHg
Diastolic Blood Pressure (DBP) | Baseline, 24 hours and 3 months after treatment
  Changes in DBP; Unit of measure: mmHg
Endothelial Function | Baseline, 24 hours and 3 months after treatment
  Measures of endothelial function taken through Flow-Mediated dilation. Unit of Measure: %

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Graziani, DDS, PhD, Principal Investigator — University of Pisa
Locations (1):
- University Hospital of Pisa, Pisa, Italy